CLINICAL TRIAL: NCT03964324
Title: Improving Diagnostics of Concurrent Inflammatory Airway Diseases in Private ENT Practice - a Study of NO Measurements in Screening for Asthma and OSA in Patients Suffering From Severe Snoring
Brief Title: NO Measurements in Screening for Asthma and OSA, in Patients With Severe Snoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christian von Buchwald (Other)
Collaborators: Bispebjerg Hospital (Other)
Responsible Party: Sponsor-Investigator, Christian von Buchwald, Clinical Professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNO07052019NOEKK
Record Dates: First submitted 2019-05-09; First posted 2019-05-28 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Snoring; Obstructive Sleep Apnea; Asthma; Airway Disease; Inflammatory Disease; Concomitant Disease
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe snorers (Experimental): Study group that will undergo fractioned exhaled nitrogen oxide measurements as well as tests of lungfunction and sleep studies. All tests are noninvasive.
  Interventions: Diagnostic Test: Fractioned Exhaled Nitrogen Oxide measurements

INTERVENTIONS:
Diagnostic Test: Fractioned Exhaled Nitrogen Oxide measurements — Measurements of Fractioned Exhaled Nitrogen Oxide obtained by blowing into a mouthpiece. The NIOX VERO machine will be used for these measures.

SUMMARY:
In Denmark an estimated 200.000 patients suffer from obstructive sleep apnoea (OSA). The breathing pauses during sleep result in varying degrees of symptoms ranging from none over disturbed sleep to severe daytime sleepiness and cognitive deficits such as reduced short-term memory and difficulty concentrating. In addition, it increases the risk of hypertension, cardiovascular thromboembolic disease and type-2 diabetes as well as causing a 3-6 times increased risk of being involved in traffic accidents.

Recent studies suggest that measurement of fractioned exhaled nitrogen oxide (FeNO) from the upper airway may be used as marker for airway inflammation. Studies have demonstrated that inflammation of the airway is present in OSA.

In this study the investigators want to see whether FeNO measurements from the upper airway can be used to screen severe snorers for OSA.

OSA is rarely diagnosed in patients with chronic rhinosinusitis (CRSwNP) or asthma. The connection between these three inflammatory conditions and the level of FeNO has not previously been investigated but might be clarified in our study.

Patients suffering from severe snoring will be offered inclusion. The patients will undergo an ENT examination as well as FeNO testing and testing of lung function. A sleep study will be made as well as they will be asked to fill out questionnaires on sleep quality, nasal symptoms, lung function and their health in general.

DETAILED DESCRIPTION:
Hypothesis FeNO can be used as screening tool for concurrent OSA and asthma in severe snorers.

Design The study is a prospective, observational multicenter trial. Patients are recruited from three different private specialist ENT-clinics where they will be offered inclusion according to guidelines. They will not be randomized and there will not be a group of patient controls.

The patients will undergo a full ENT-examination including a fiberoptic examination of both nasal cavities and the upper airway. NO-measurements as well as tests of lung function and sleep studies (Cardio-Respiratory-Monitoring = CRM) will also be performed. Furthermore, patients will be asked to fill out three questionnaires (see below). Patients with severe snoring and mild OSA will be offered an evaluation and a DISE (Drug Induced Sedation Endoscopy) at the ENT department Rigshospitalet, Gentofte.

NO-measurements:

FeNO-measurements will be carried out using a handheld NO-device (NIOX VERO, Aerocrine AB, Solna, Sweden). The patients will be asked to blow into a mouthpiece on the device which will then calculate the level of FeNO.

Lung function:

Tests of lung function will be carried out using EasyOne Pulmonary Function Device where the patients will blow into a mouthpiece.

Sleep studies:

Sleep studies (Cardio-Respiratory Monitoring = CRM) will be done as overnight home-studies using SOMNOtouch RESP that will measure heartrate, oxygen saturation, movement of chest and abdomen. All measurements are non-invasive.

Questionnaires:

Patients will be asked to fill out questionnaires regarding nasal symptoms (Sino-Nasal Outcome Test = SNOT-22) along with questionnaires on sleep quality (Epworth Sleepiness Scale = ESS), lung function (ACQ) and general health (The Danish version of Short Form (SF-36) Health Survey) developed at RAND as part of the Medical Outcomes Study (MOS). Danish validated version by Bjørner JB et al.

Statistics Data will be processed using IBM SPSS (Chicago, USA). For categorical data Pearson's Chi2-test or Fischer's exact tests will be used. Students T-test for normally distributed data, while data that are not normally distributed will be analyzed using Mann Whitney U-test. Shapiro-Wilks test or graphic plots will be used in the evaluation of data distribution.

Calculation of Power:

FeNO levels in simple snorers compared to snorers with concurrent asthma or OSA.

Expected incidence of a severe snorer also having OSA: 25% Expected incidence of OSA in the general adult population: 10% Power: 0.8 Significance: 0.5 Sample size: 40 severe snorers

Risks, disadvantages and advantages:

There are no known risks associated with the tests of lung function or FeNO measurements. A bit of discomfort with blowing forcefully into the mouthpieces during the tests might occur. The fiberoptic examination of the upper airway might also result in a bit of discomfort. It is expected that paracetamol is sufficient treatment. In the unlikely case that paracetamol is not enough patients will be instructed to contact their physician.

Inclusion in the study will provide the patients with a very thorough examination illuminating any concurrent diseases that might explain their symptoms and discomfort. If any concurrent disease is found, they will be referred for further specialist treatment.

Safety precautions The patients will all be examined by specialists in ENT, who are used to performing these examinations. All will be thoroughly informed about the tests and the motivation for performing them.

In the unlikely event of pronounced discomfort during a test, it will be stopped.

Biobank No tissue samples will be collected.

Data from patient files The investigators have requested access to the patient files in the local IT-systems in the three private ENT clinics as well as via Sundhedsplatformen and FMK (Fælles Medicin Kort) to verify any medical treatment that might interfere with the study as stated in the inclusion and exclusion criteria.

Prior to inclusion, and consent to participate in the study, data on age, previous illness, current medication, and results from the ear-nose-and throat examination will be requested, in order to verify that the participants are eligible for inclusion. The information will be passed on to the investigators.

After inclusion and consent is given to participate in the study, data on allergies, weight, height, age, gender, concurrent illness, and current medication, will be requested.

Consent to participate in the study allows the investigators, sponsors, representatives of sponsors, as well as the supervisory, direct access to collection of data from patient files, including the electronic files, to get information on health-related issues necessary to conduct the research project, self-monitoring, and quality-monitoring, as obligated.

Handling of personal data:

The rules of Databeskyttelsesordningen / persondataforordning will be followed. Data will be stored in accordance with guidelines and only after approval from the local Data Protection Agency (Datatilsynet).

Responsibility for data:

A: Key investigator Eva Kirkegaard Kiær M.D., ENT-specialist Department of otorhinolaryngology, Head and Neck Surgery and Audiology Rigshospitalet, Copenhagen University Hospital Blegdamsvej 9, 2100 København Ø

+ 45 35 45 66 35 / 26 70 17 10 eva.kirkegaard.kiaer.01@regionh.dk

B: Investigator Christian von Buchwald M.D., D.M.Sci Department of otorhinolaryngology, Head and Neck Surgery and Audiology Rigshospitalet, Copenhagen University Hospital Blegdamsvej 9, 2100 København Ø

+ 45 35 45 20 70 christian.von.buchwald@regionh.dk

C: Investigator Nina Vibeke Backer M.D., D.M.Sci Department of Respiratory Medicine Bispebjerg Hospital Ebba Lunds Vej 48, 2400 København NV + 45 38 63 51 22 backer@dadlnet.dk

D: Investigator Andreas Tomaas Ravn M.D., ENT-specialist Frederiksberg øre-næse-halsklinik Falkoner Allé 15, 1. tv., 2000 Frederiksberg + 45 38 87 84 98 atravn@hotmail.com

E: Investigator Steffen Ørntoft M.D., ENT-specialist Øre Næse Hals Klinikken Gammel Køge Landevej 263 1. th., 2650 Hvidovre

+ 45 36 78 88 03 orntoft@dadlnet.dk

F: Investigator Christian Prætorius and Roland Welinder M.D., ENT-specialists Øre-næse-halsklinikken i Hørsholm Kongevejscentret 6, 1. Sal, 2970 Hørsholm

+ 45 45 86 46 00 chr.praetorius@dadlnet.dk

Key investigator is responsible for the safe storage of data in accordance with the guidelines from the local Data Protection Agency (Datatilsynet). Patient data will be stored in a locked cabinet in a locked office.

In accordance with the Danish Law on Health §46, 1+3, the same group of physicians will collect data, process data and publish data. Only investigators A, B and C will process data.

Initiative The initiative for the study is a collaboration between investigator A, B, C and D. All the aforementioned investigators have contributed to the outlines of the study.

Funding The study is partially funded by Fonden for Faglig Udvikling i Speciallægepraksis (FAPS) and Øre-næse-halskirurgisk og Audiologisk Klinik, Rigshospitalet.

All the funding is managed by a research account at Rigshospitalet. The key investigator is employed by the Øre-næse-halskirurgisk and Audiologisk Klinik, Rigshospitalet, but does not have a financial association to FAPS.

Remuneration The patients will not be offered remuneration.

Recruitment Patients will be recruited from three private ENT clinics (investigators D-F). Patients will make appointments for consultation in the clinics as usual, based on their symptoms, and will be offered inclusion in the study if they fall under the inclusion criteria and not the exclusion criteria. All will have the opportunity to consider inclusion in the study and will be offered a new consultation if needed.

Information In accordance with guidelines from the Ethics Committee, participating patients will be given both written and oral information about the study, purpose, and consequences. Patients will receive the folder "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt Forskningsprojekt" published by National Videnskabsetisk Komité (the Central Ethics Committee).

When considering inclusion in the study patients will be offered a new consultation where they can bring an assessor. There will be time and opportunity for any questions they might have. It will take place in an undisturbed location as to ensure a comfortable environment for conversation. Patients will be informed that participation is optional, and their treatment will not be affected should they choose not to accept inclusion.

Patients will be informed of their right to decline information on essential health related issues. The informing physician is responsible for ensuring that the information is understood. The patient has the right to a minimum of one week to consider inclusion.

Informed consent On the day of inclusion, or no later than 14 days after, a written consent will be obtained. The investigator signs the informed consent stating that the patient has received both written and oral information about the project.

Patients will be informed that they can withdraw their informed consent at any given time, and that it will not affect any current or future treatment or consultation.

Should any essential information about a patient's health appear during the study they will be informed accordingly, unless they have clearly stated that they decline such information.

Publication When the results of the study are available, one of the physicians (A-F) will, as far as possible, inform the patients in the study. Information regarding patients is protected by "Lov om behandling af personoplysninger" and "Lov om patienters retstilling (sundhedsloven afsnit III)".

Results, both positive, negative or inconclusive, will be published after the completion of the study. If publication in a peer review journal is not possible, results will be published through other media channels. The study will be registered at www.clinicaltrials.gov

Ethical considerations The study is approved by the local Ethics Committee as well as the Data Protection Agency The purpose of the study is to improve treatment of patients with CRSwNP by diagnosing other conditions that might affect their treatment and quality of life if undiagnosed. The conditions of interest (OSA and asthma) have symptoms that mimic CRSwNP and can therefore be difficult to diagnose if one is not careful to look for them. With this study the investigators hope to find a simple test, associated with minimal discomfort, that might help screen these patients for OSA and asthma.

OSA and asthma are conditions associated with severe consequences on both quality of life and comorbidity. Hopefully a quick diagnosis will help the patients to relevant treatment thus reducing their risk of long-term sequelae.

Any discomfort during the study seems minimal in contrast to the health benefits it will grant patients that are diagnosed with comorbidity as OSA and asthma.

Insurance Patients are covered by "patienterstatningen" during the study period.

ELIGIBILITY:
Inclusion Criteria:

• Severe snorers that seek help based on their personal health and/or social limitations due to their snoring.

Exclusion Criteria:

* Patients with known OSA
* Patients with nasal polyps
* Other inflammatory diseases of the upper airways (i.e. cystic fibrosis, primary ciliary dyskinesis) or immune deficiencies, sarcoidosis or systemic vasculitis
* Infections in the upper airway during the past two weeks
* Smokers
* Treatment with antidepressant or sedative drugs
* Age below 18
* Patients unable to give an informed consent
* Patients that do not speak or read Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Fractioned Exhaled Nitric Oxide (FeNO) | 3 years
  Fractioned exhaled nitric oxide (FeNO) parts per billion (ppb) will be measured at an exhalation flow rate of 0.05 L/s, during single exhalation, using a portable nitric oxide analyzer device (NIOX VERO, Circassia AB, P.O. Box 3006 SE-750 03 Uppsala, Sweden). The normal exhaled NO values during measurements will be set to 5-35 ppb for healthy adults. Patients must produce a 10-second exhalation of breath at an exhalation pressure of 10-20 cmH2O to maintain a stable flow rate of 50±5 mL/s. A calibrated electrochemical sensor evaluates the final 3 seconds of exhalation expressing results in ppb with a range between 5 ppb and 300 ppb. The higher the measurement the larger is the risk of airway inflammation.

SECONDARY OUTCOMES:
Nasal Nitric Oxide (nNO) | 3 years
  Nasal Nitric Oxide (nNO) parts per billion (ppb) will be measured both as tidal breathing (TB-nNO) and as expiration against resistance (ER-nNO). A portable nitric oxide analyzer device (NIOX VERO, Circassia AB, Uppsala, Sweden) will be used for all nNO´s.
  TB-nNO is a measurement of the level of nitric oxide from one side of the nose as the patient breathes through the open mouth. The device will collect data for 30 s. Results vary in ppb from 5-1500 (580 is the mean for healthy subjects).
  ER-nNO will be performed while the patient breathes through the mouth against a restrictor (mouthpiece). After a complete inhalation to the full capacity of the lungs the patient will exhale against the restrictor with the lips closed around the mouthpiece. The patient should exhale steadily for 30 s as the device measures nitric oxide from one side of the nose. Results vary in ppb from 5-1500 with (915 is the mean for healthy subjects).
Forced Expiratory Volume in 1 second (FEV1) | 3 years
  Spirometry will be performed using MiniSpir Spiro (Alere A/S Denmark). With a nose clip on the nose patients will be instructed to exhale into a mouthpiece after inhalation to full capacity of the lungs.
  The FEV1 (forced expiratory volume in 1 s) is the volume exhaled during the 1st second of a forced exhalation measured in liters. Values below 80 % of the expected normal value, matched by age and height, is considered significantly reduced. The normal value for a 175 cm tall and 50-year-old male is 3,50 L. The normal value for a similar female is 2,99 L.
Apnea Hypopnea Index (AHI) | 3 years
  Cardio Respiratory Monitoring (CRM) will be performed using SOMNOtouch RESP. As an overnight home-study the equipment will measure flow of air and snoring using a nasal cannula. Puls rate, oxygen saturation and heartrate will be measured as well as movement of the thorax and abdomen and body position. Based on these registrations the system will calculate an AHI (apnea-hypopnea index). This index is the average sum of apneas and hypopneas per hour of sleep. An apnea is a full cessation of breathing for a minimum of 10 s followed by a desaturation of at least 3%. A hypopnea is a 50% or larger reduction in breathing for a minimum of 10s. An index below 5 is normal. An index above 5 is diagnostic of obstructive sleep apnea.
Sino Nasal Outcome Test (questionnaire) | 3 years
  SNOT-22 (Sino Nasal Outcome Test). 22 questions on sino nasal symptoms. Answers rank from 0-5 where 0 is "not a problem" and 5 is "worst possible problem". Total scores range from 0-110.
ESS (questionnaire) | 3 years
  ESS (Epworth Sleepiness Scale). 8 questions on daytime sleepiness in every-day situations. Answers rank from 0-3 where 0 is "not a problem" and 3 is "would fall asleep". Total scores range from 0-24. A score higher than 9 is considered excessive daytime sleepiness and indicates a risk of having obstructive sleep apnea.
Short Form 36 questionnaire | 3 years
  The SF-36 questionnaire (Short Form 36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 is a measure of health status. The original SF-36 stemmed from the Medical Outcome Study, MOS, which was conducted by the RAND Corporation.
  The questionnaire of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. The scores are calculated using special software.
ACQ (questionnaire) | 3 years
  ACQ (asthma control questionnaire). The ACQ has 7 questions. Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). Clinic staff score the FEV1% predicted on a 7-point scale. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
  The ACQ can identify the adequacy of asthma control in individual patients. In general, patients with a score below 1.0 will have adequately controlled asthma and above 1.0 their asthma will not be well controlled.

CONTACTS AND LOCATIONS:
Overall Officials: Eva K Kiaer, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- University Hospital of Copenhagen, Rigshospitalet, Copenhagen, Capital Region, Denmark

REFERENCES:
- [Derived] Kiaer E, Ravn A, Jennum P, Praetorius C, Welinder R, Orntoft S, von Buchwald C, Backer V. Fractional exhaled nitric oxide-a possible biomarker for risk of obstructive sleep apnea in snorers. J Clin Sleep Med. 2024 Jan 1;20(1):85-92. doi: 10.5664/jcsm.10802. PMID 37707290